CLINICAL TRIAL: NCT02094924
Title: An Open-Label, Randomised, Single Dose, Two-Way Crossover Pilot Study to Determine the Relative Bioavailability of a Fixed Dose Combination Tablet Formulation of GSK587323 (16mg Candesartan Cilexetil/12.5mg Hydrochlorothiazide) Relative to Respective Reference Dosage Atacand D in Healthy Adult Human Subjects Under Fasting Conditions
Brief Title: A Relative Bioavailability Study of a Fixed Dose Combination (FDC) Tablets of GSK587323
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200957
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
Keywords: Candesartan cilexetil; Hypertension; Hydrochlorothiazide; Healthy adult human subjects; Bioequivalence
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Participants in this arm will receive treatment A in period 1 and treatment B in period 2. Subjects will receive a single reference FDC tablet of 16mg candesartan cilexetil/12.5mg HCTZ as Treatment A administered orally with 240mL of water and a single 16mg candesartan cilexetil/12.5mg HCTZ FDC tablet (GSK587323) as Treatment B.
  Interventions: Drug: GSK587323; Drug: FDC of candesartan cilexetil 16 mg and HCTZ 12.5mg
- Sequence 2 (Experimental): Participants in this arm will receive treatment B in period 1 and treatment A in period 2. Subjects will receive a single reference FDC tablet of 16mg candesartan cilexetil/12.5mg HCTZ as Treatment A administered orally with 240mL of water and a single 16mg candesartan cilexetil/12.5mg HCTZ FDC tablet (GSK587323) as Treatment B.
  Interventions: Drug: GSK587323; Drug: FDC of candesartan cilexetil 16 mg and HCTZ 12.5mg

INTERVENTIONS:
Drug: GSK587323 — Single dose of FDC tablet formulation to be taken orally.
Drug: FDC of candesartan cilexetil 16 mg and HCTZ 12.5mg — Single dose of FDC tablet formulation to be taken orally

SUMMARY:
This study is required to confirm the suitability of a candidate FDC of 16mg candesartan cilexetil/12.5mg HCTZ (GSK587323) formulation for further development and provide data to allow the design of a future pivotal bioequivalence study. This study aims to determine the relative bioavailability of a FDC tablet formulation of 16mg candesartan cilexetil/12.5mg HCTZ relative to the reference product of same fixed dose combination (16mg candesartan cilexetil/12.5mg HCTZ) in healthy adult humans. This will be an open-label, randomised, single dose, two-way crossover study. Each subject will participate in two treatment periods and will be randomized to one of two sequences and administered one of the two treatments, A or B, as per the randomization schedule. The two treatment periods will be separated by a washout period of 7 to 14 days to ensure the candesartan and HCTZ have been effectively eliminated from the subject between dosing occasions. The study will enroll 16 healthy subjects to ensure that 14 subjects complete the study as planned.

ELIGIBILITY:
Inclusion Criteria:

* Subjects Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Male and females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the GlaxoSmithKline (GSK) Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50kilograms (kg) and Body Mass Index (BMI) within the range 19 - 24.9kg / meter^2 (m^2) (inclusive).
* A female subject is eligible to participate if she is of: non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records; or postmenopausal defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli international units per millilitre (MlU/mL) and estradiol < 40 picograms per millilitre (pg/mL) (<147 picomol per litre (pmol/L)) is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* A female subject is eligible to participate if she is of child-bearing potential with negative pregnancy test as determined by serum or urine Human Chorionic Gonadotropin (hCG) test at screening or prior to dosing AND agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up contact visit.
* A female subject is eligible to participate if she has only same-sex partners, when this is her preferred and usual lifestyle.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods. This criterion must be followed from the time of the first dose of study medication until the follow-up contact visit.
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin 1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single or averaged QT duration corrected for heart rate (QTc) of triplicate Electrocardiograms (ECGs) obtained over a brief recording period: QT duration corrected for heart rate by Fridericia's Formula (QTcF) < 450 millisecond (msec).

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Gastrointestinal disease or with gastrointestinal surgical history which can affect the absorption of the investigational drug.
* Any subject with a systolic blood pressure (BP)<95 millimetre of Mercury (mmHg) or with a recent history of postural symptoms
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04-17 (Actual); Primary Completion 2014-05-23 (Actual); Study Completion 2014-05-23 (Actual)

PRIMARY OUTCOMES:
Composite of PK parameters for candesartan and HCTZ to assess relative bioavailability. | Pre dose, 0.33, 0.67, 1, 1.33, 1.67, 2.0, 2.33, 2.67, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 10, 12, 16, 24, 36, and 48hours post dose in each treatment period.
  PK parameters include: maximum observed plasma concentration (Cmax), area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC [0-infinite]) and area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments (AUC [0-t]). Twenty four blood samples (1x 5mililiter (mL)) will be collected at the specified time points for PK analysis of candesartan and HCTZ.

SECONDARY OUTCOMES:
PK profile of candesartan and HCTZ. | Pre dose, 0.33, 0.67, 1, 1.33, 1.67, 2.0, 2.33, 2.67, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 10, 12, 16, 24, 36, and 48hours post dose in each treatment period.
  PK parameters included: time to Cmax (tmax), Percentage of AUC (0-infinite) obtained by extrapolation, and apparent terminal phase half-life (t1/2). PK blood samples (1x 5mL)) will be collected at the specified time points for PK analysis of candesartan and HCTZ.
Vital sign assessment as a measure of safety and tolerability. | Up to 39 days
  Vital sign parameters include: systolic blood pressure, diastolic blood pressure, and pulse rate. At Baseline the average of the last two blood pressures and pulse readings will be recorded. All measurements will be measured in supine position after 5 minutes rest.
Review of adverse events (AEs) as a measure of safety and tolerability. | Up to 39 days
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. All AEs and serious AEs (SAEs) will be collected from the start of dosing with Investigational Product and until the follow-up visit. However, any SAEs related to study participation or concomitant
Clinical laboratory data assessment as measure of safety and tolerability. | Up to 39 days
  All subjects for all treatments will be evaluated for any abnormal laboratory test results (haematology, clinical chemistry, or urinalysis).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hyderabad, India

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 200957 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/200957?search=study&search_terms=200957#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 200957 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200957 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200957 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200957 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200957 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200957 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200957 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register